CLINICAL TRIAL: NCT07162675
Title: A Multicenter Prospective Study: The Impact of Step Count Measured by Smartwatches on Treatment Response in Non-Metastatic HER2-Negative Breast Cancer Patients Receiving Neoadjuvant Therapy
Brief Title: Step Count and Treatment Response in Neoadjuvant Breast Cancer
Acronym: NEOBRE-STEP
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK2-2025-454; AEŞH-BADEK2-2025-454 (Other: Ankara Etlik City Hospital Scientific Research Ethics Committee)
Record Dates: First submitted 2025-08-24; First posted 2025-09-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm Malignant Female; Exercise; Breast Cancer Females; Wearable Technology; Sleep Quality; Smartwatches
Keywords: neoadjuvant therapy; HER2-Negative Breast Cancer; Smartwatch; Step Count; Physical Activity; Patient-Reported Outcomes; Quality of Life (EORTC QLQ-C30)
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant HER2-Negative Breast Cancer Patients: This cohort includes female patients aged ≥18 years with non-metastatic, HER2-negative breast cancer who are scheduled to receive neoadjuvant systemic therapy followed by surgery.
  Interventions: Device: Huawei Fit 2 Smartwatch

INTERVENTIONS:
Device: Huawei Fit 2 Smartwatch — Participants will receive a Huawei Fit 2 smartwatch within the first week of initiating neoadjuvant systemic therapy. The device will be worn throughout the treatment period to continuously monitor step counts, physical activity intensity, sleep duration, and heart rate. It is used solely for non-invasive monitoring and does not alter the standard oncological treatment.

SUMMARY:
This prospective multicenter observational study (NEOBRE-STEP) investigates the impact of daily step counts, measured by Huawei Fit 2 smartwatches, on treatment response in patients with non-metastatic Human Epidermal Growth Factor Receptor 2 (HER2)-negative breast cancer undergoing neoadjuvant systemic therapy. Patients will wear smartwatches to continuously record step counts, activity intensity, sleep, and heart rate. Patient-reported outcomes, including sleep quality (Pittsburgh Sleep Quality Index, PSQI) and quality of life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30, EORTC QLQ-C30), will be assessed at baseline and after treatment. The primary outcomes are pathological complete response (pCR) and Miller-Payne score. Secondary outcomes include sleep quality, quality of life, perioperative outcomes, and feasibility of smartwatch monitoring.

DETAILED DESCRIPTION:
Physical activity and sleep quality are important prognostic factors in oncology, but objective and continuous monitoring during neoadjuvant systemic therapy is limited. Wearable devices provide non-invasive, real-time data on step counts, heart rate, and sleep. This study will evaluate whether daily step counts and digital health metrics predict pathological response in non-metastatic Human Epidermal Growth Factor Receptor 2 (HER2)-negative breast cancer.

Primary Objective: To assess the association between daily step counts and pathological response, including pathological complete response (pCR, defined as no residual invasive carcinoma in the breast and axillary nodes) and Miller-Payne score (range 1-5; higher scores indicate greater regression).

Secondary Objectives: To explore associations between physical activity and sleep quality (Pittsburgh Sleep Quality Index, PSQI), quality of life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30, EORTC QLQ-C30), and perioperative outcomes; and to evaluate feasibility and adherence to smartwatch monitoring.

Methods: This is a multicenter prospective observational cohort study enrolling 82 female patients aged ≥18 years with non-metastatic HER2-negative breast cancer scheduled to receive neoadjuvant systemic therapy followed by surgery. Smartwatches (Huawei Fit 2) will continuously monitor activity, sleep, and heart rate. Questionnaires will be administered at baseline and at the end of treatment.

PSQI: Global score 0-21; higher scores indicate worse sleep quality; a cut-off >5 defines poor sleep. A validated Turkish version is available.

EORTC QLQ-C30: Standardized 0-100 scoring system; higher scores on functional scales indicate better functioning, while higher scores on symptom scales indicate greater symptom burden. A validated Turkish version is available.

Pathological response will be determined at surgery using pCR and Miller-Payne criteria.

Sample Size and Statistics: A priori power analysis (effect size d = 0.5, α = 0.05, power = 0.80) indicates a minimum of 82 patients. Regression analyses and subgroup evaluations will test associations with step counts, questionnaire scores, and perioperative outcomes.

Significance: This study (NEOBRE-STEP) is among the first multicenter efforts to integrate wearable health monitoring into breast cancer supportive care. By combining objective activity and sleep data with validated patient-reported outcomes, the study may provide new prognostic insights and support the integration of digital health tools into oncology practice.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.
* Pathologically confirmed non-metastatic HER2-negative breast cancer.
* Candidates scheduled to receive neoadjuvant systemic therapy followed by surgery.
* ECOG performance status 0-2.
* Ability to provide informed consent.

Exclusion Criteria:

* Metastatic breast cancer at diagnosis.
* HER2-positive breast cancer.
* Previous systemic therapy for current breast cancer.
* Severe comorbidities limiting mobility or physical activity (e.g., advanced neurologic or musculoskeletal disorders).
* ECOG performance status ≥3.
* Pregnancy or breastfeeding.
* Refusal or inability to use a smartwatch device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biologically female patients with pathologically confirmed non-metastatic HER2-negative breast cancer are eligible for participation.
Study Population: The study population will consist of eighty-two female patients with non-metastatic, HER2-negative breast cancer who are scheduled to receive neoadjuvant systemic therapy followed by surgery. All participants will be recruited consecutively from the Department of Medical Oncology at Ankara Etlik City Hospital and Gazi University Faculty of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | From initiation of neoadjuvant therapy to the date of surgery (expected range: 24-32 weeks after treatment initiation).
  Defined as the absence of residual invasive carcinoma in the breast and axillary lymph nodes at surgery. Pathological response will be evaluated after completion of neoadjuvant systemic therapy.
Miller-Payne Tumor Regression Score | From initiation of neoadjuvant therapy to the date of surgery (expected range: 24-32 weeks after treatment initiation).
  Histopathological regression grading system ranging from 1 (minimal regression) to 5 (complete disappearance of invasive cancer). Higher scores indicate greater regression.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) Score | Baseline (within first week of therapy) to completion of neoadjuvant therapy (24-32 weeks).
  Patient-reported questionnaire assessing global sleep quality. Score range: 0-21; higher scores indicate worse sleep quality. A cut-off >5 defines poor sleep quality. A validated Turkish version is available.
EORTC QLQ-C30 Global Health and Functional Scales | From baseline (within first week of neoadjuvant therapy) to completion of neoadjuvant therapy (24-32 weeks).
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30. Scores standardized to 0-100. Higher scores on functional scales represent better functioning; higher scores on symptom scales represent worse symptom burden. A validated Turkish version is available.

OTHER OUTCOMES:
Device-Measured Physical Activity Intensity | From treatment initiation to end of neoadjuvant therapy (up to 32 weeks).
  Minutes per day spent in moderate-to-vigorous physical activity, including bouts ≥10 minutes, measured by smartwatch.
Resting Heart Rate (RHR) | From treatment initiation to end of neoadjuvant therapy (up to 32 weeks).
  Average weekly resting heart rate measured by smartwatch (beats per minute). Changes from baseline will be evaluated.
Device-Measured Sleep Duration | From device allocation to end of neoadjuvant therapy (up to 32 weeks).
  Nightly sleep duration derived from smartwatch recordings, measured in hours per night.
Device-Measured Sleep Efficiency | From device allocation to end of neoadjuvant therapy (up to 32 weeks).
  Proportion of time asleep relative to time in bed, derived from smartwatch recordings, expressed as percentage (%).
Correlation Between Device-Measured Sleep Duration and PSQI Score | From device allocation to end of neoadjuvant therapy (up to 32 weeks).
  Statistical correlation between nightly sleep duration and PSQI scores.
Correlation Between Device-Measured Sleep Efficiency and Miller-Payne Score | From device allocation to surgery (up to 32 weeks).
  Statistical correlation between sleep efficiency and histopathological regression grading.
Correlation Between Device-Measured Sleep Efficiency and PSQI Score | From device allocation to end of neoadjuvant therapy (up to 32 weeks).
  Statistical correlation between sleep efficiency and PSQI scores.
Correlation Between Device-Measured Sleep Duration and Miller-Payne Score | From device allocation to surgery (up to 32 weeks).
  Statistical correlation between nightly sleep duration and histopathological regression grading.
Correlation Between Device-Measured Sleep Duration and Pathological Complete Response (pCR) | From device allocation to surgery (up to 32 weeks).
  Statistical correlation between nightly sleep duration and pathological complete response status.
Correlation Between Device-Measured Sleep Efficiency and Pathological Complete Response (pCR) | From device allocation to surgery (up to 32 weeks).
  Statistical correlation between sleep efficiency and pathological complete response status.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Ankara Etlik City Hospital; Orhun Akdoğan, MD, Principal Investigator — Gazi University Medical Oncology Departmant, Ankara
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Medical Oncology Department, Ankara, Yenimahalle
  - Gazi University Medical Oncology Department, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No